CLINICAL TRIAL: NCT02438891
Title: Treatment of Tinnitus Using a Web-based Sound and Cognitive Behavioral Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Hamid Djalilian, Director, Division of Neurotology and Skull Base Surgery, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-1358
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBT course (Experimental): 8-week internet-based cognitive behavioral therapy and sound therapy course
  Interventions: Behavioral: Cognitive behavioral therapy

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — Cognitive behavioral therapy is a form of tinnitus psychotherapy which aims to help patients control negative thoughts or emotions associated with tinnitus.

SUMMARY:
Most tinnitus sufferers experiences significant anxiety or depression that worsens the subjective symptoms related to tinnitus. In this study, we intend to use internet-based cognitive behavioral therapy (CBT) in addition to sound therapy to provide psychotherapy to patients with tinnitus. Multiple research studies have found CBT to be effective in improving the subjective symptoms of tinnitus. The internet-based CBT course developed for this study is 8 weeks in duration and organized into eight 1-week modules; each module contains 2-4 separate lessons and homework assignments. Patients will be given unique usernames and passwords. In each weekly module, patients will review educational materials online, do exercises. and will be given feedback based on the results of the completed exercises. In addition, patients are given different meditation exercises each week for relaxation and coping with their tinnitus. These interactive materials enable patients to manage and control any negative feelings and thoughts that may be associated with tinnitus and help take their attention away from tinnitus. Tinnitus loudness and annoyance will be measured before and after the program. An internet-based course enables care providers to monitor patients' progress with the CBT course remotely, and allows patients to learn CBT at their own convenience and schedule.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate a internet-based cognitive behavioral therapy (CBT) system as a method of treating patients with tinnitus. Tinnitus is a common symptom that is defined as the perception of the sound in the ears without any external source. It is often described by the patients as ringing or a buzzing sound, alone or more often as a mixture of sounds. This symptom afflicts 10 to 15% of the adult population. It usually does not bother patients significantly; however about 10% of the patients will suffer severe problems which include insomnia, anxiety, depression and other emotional problems. The various forms of treatment for tinnitus that have been tested in properly controlled trials can be classified as pharmacological, sound therapy and psychological. In clinical trials, no pharmacological agent has been shown to have lasting effect on the presence or severity of tinnitus. Despite numerous available treatments for tinnitus, it is rarely curable and the sufferer must use coping strategies to decrease the distress.

CBT is a psychological treatment that has emerged as consistently beneficial in terms of affecting overall well-being and reducing the level of tinnitus-related annoyance. CBT is a form of psychotherapy for tinnitus that intends to measure and improve the affected individual's reaction to tinnitus. It does not eliminate the auditory perception, but reduces or corrects negative responses to tinnitus. CBT identifies negative automatic thought and determines its validity with the patient. It intends to modify negative automatic thoughts to more positive and realistic ones. Using this method, the patients with tinnitus can function better despite the presence of tinnitus.

One of the problems with CBT is the shortage of clinicians who are specialized in CBT for tinnitus. For this reason, some programs have been developed which utilize guided or therapist-supported self-help approach. Internet based CBT have been developed for patients with tinnitus in several studies. Anderson and colleagues in Sweden compared pre and post therapeutic effect of CBT in 117 participants with tinnitus duration of more than 6 months. All subjects had been offered the CBT program and 96 provided outcome measures. Tinnitus-related distress, depression, and diary ratings of annoyance decreased significantly. Also in comparison to a control group, they found out that these patients showed an improvement of at least 50% on the Tinnitus Reaction Questionnaire. They concluded that CBT via the Internet can help individuals decrease annoyance associated with tinnitus. In another study by Kaldo et.al., they evaluated the difference between internet-based CBT and group-based CBT. The subjects in internet treatment consumed less therapist time and it was 1.7 times as cost-effective as the group treatment. However some studies support the utilization of self-help methods for treatment of tinnitus, but there are still some problems with using these methods such as accessibility to internet, knowledge of the patients on using computers and internet, interactivity and user friendly structure of the software that is used for the program and time management of the patients for practicing methods and exercises embedded in this program. By correcting and rectifying these 3 of 25 issues, internet-based self-help programs will better serve the patients with their cost-effective and time saving benefits. Currently there is no web-based CBT for the treatment of tinnitus available.

The objective of this study is to evaluate an internet-based CBT course for the treatment of tinnitus. Adult patients (18+ years) with moderate-to-severe tinnitus (see additional Inclusion Criteria) will be selected for enrollment and will take pre-course surveys and undergo tinnitus-specific audiometry testing. The 8-week course will be completed by the patients online, at home. Following completion of the course, enrollees will repeat the surveys and tinnitus-specific audiometry tests.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with the chief complaint of tinnitus for 6 months or more
2. 18 years or older
3. Male or Female
4. Internet and e-mail access at home
5. Adequate command of English to fill out the surveys and questionnaires in the website

Exclusion Criteria:

1. Aged less than 18 years
2. History of Psychosis
3. Subjects currently taking medications known to cause tinnitus (aspirin, ibuprofen, naproxen) which cannot be stopped.
4. Active illicit drug use, alcohol dependence
5. Patients with severe depression based on the Beck's depression inventory survey scores
6. Patients with severe anxiety based on the GAD-7 survey scores
7. Patients with severe Post Traumatic Stress Disorder (PTSD) based on the PTSD- civilian version survey
8. Not currently undergoing CBT with a Psychologist
9. No other concurrent tinnitus therapy
10. Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-07-14 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2020-12-16 (Actual)

PRIMARY OUTCOMES:
Subjective improvement of tinnitus | 9 weeks
  Subjective improvement, from baseline, of tinnitus-related stress, emotions, feelings and thoughts. Evaluated by pre- and post-course audiometry and surveys, and patient feedback.

SECONDARY OUTCOMES:
Beck's depression survey | 9 weeks
  pre-course and post-course survey for subjective assessment of tinnitus
Post-traumatic Stress Disorder civilian survey | 9 weeks
  pre-course and post-course survey for subjective assessment of tinnitus
Tinnitus handicap inventory survey | 9 weeks
  pre-course and post-course survey for subjective assessment of tinnitus
GAD-7 survey | 9 weeks
  pre-course and post-course survey for subjective assessment of tinnitus

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Djalilian, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California Irvine Medical Center, Orange, California, United States

REFERENCES:
- [Background] Cima RF, Maes IH, Joore MA, Scheyen DJ, El Refaie A, Baguley DM, Anteunis LJ, van Breukelen GJ, Vlaeyen JW. Specialised treatment based on cognitive behaviour therapy versus usual care for tinnitus: a randomised controlled trial. Lancet. 2012 May 26;379(9830):1951-9. doi: 10.1016/S0140-6736(12)60469-3. PMID 22633033
- [Background] Zachriat C, Kroner-Herwig B. Treating chronic tinnitus: comparison of cognitive-behavioural and habituation-based treatments. Cogn Behav Ther. 2004;33(4):187-98. doi: 10.1080/16506070410029568. PMID 15625793
- [Background] Andersson G, Kaldo V. Internet-based cognitive behavioral therapy for tinnitus. J Clin Psychol. 2004 Feb;60(2):171-8. doi: 10.1002/jclp.10243. PMID 14724924
- [Background] Sweetow RW. Cognitive aspects of tinnitus patient management. Ear Hear. 1986 Dec;7(6):390-6. doi: 10.1097/00003446-198612000-00008. PMID 3792682
- [Result] Jasper K, Weise C, Conrad I, Andersson G, Hiller W, Kleinstauber M. Internet-based guided self-help versus group cognitive behavioral therapy for chronic tinnitus: a randomized controlled trial. Psychother Psychosom. 2014;83(4):234-46. doi: 10.1159/000360705. Epub 2014 Jun 19. PMID 24970708
- [Result] Kaldo V, Haak T, Buhrman M, Alfonsson S, Larsen HC, Andersson G. Internet-based cognitive behaviour therapy for tinnitus patients delivered in a regular clinical setting: outcome and analysis of treatment dropout. Cogn Behav Ther. 2013;42(2):146-58. doi: 10.1080/16506073.2013.769622. Epub 2013 Feb 25. PMID 23432207
- [Result] Hesser H, Gustafsson T, Lunden C, Henrikson O, Fattahi K, Johnsson E, Zetterqvist Westin V, Carlbring P, Maki-Torkko E, Kaldo V, Andersson G. A randomized controlled trial of Internet-delivered cognitive behavior therapy and acceptance and commitment therapy in the treatment of tinnitus. J Consult Clin Psychol. 2012 Aug;80(4):649-61. doi: 10.1037/a0027021. Epub 2012 Jan 16. PMID 22250855
- [Result] Kaldo V, Levin S, Widarsson J, Buhrman M, Larsen HC, Andersson G. Internet versus group cognitive-behavioral treatment of distress associated with tinnitus: a randomized controlled trial. Behav Ther. 2008 Dec;39(4):348-59. doi: 10.1016/j.beth.2007.10.003. Epub 2008 Apr 20. PMID 19027431
- [Result] Kaldo-Sandstrom V, Larsen HC, Andersson G. Internet-based cognitive-behavioral self-help treatment of tinnitus: clinical effectiveness and predictors of outcome. Am J Audiol. 2004 Dec;13(2):185-92. doi: 10.1044/1059-0889(2004/023). PMID 15903144